CLINICAL TRIAL: NCT00535132
Title: A Blinded-initiation Study of Medication Satisfaction in Subjects With Schizophrenia Treated With Paliperidone ER After Suboptimal Response to Oral Risperidone
Brief Title: Study to Measure Drug Satisfaction of Patients With Schizophrenia After Switching From Risperidone to Paliperidone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014347; R076477SCH4013
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2009-10-20 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; medication satisfaction, Invega
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 002 (Experimental): Oral Risperidone 4 or 6 mg MG once daily for 0-2 weeks
  Interventions: Drug: Oral Risperidone
- 001 (Experimental): Paliperidone ER 6, 9 or 12 MG once daily for 4-6 weeks
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Oral Risperidone — 4 or 6 mg MG once daily for 0-2 weeks
  Arms: 002
Drug: Paliperidone ER — 6, 9 or 12 MG once daily for 4-6 weeks
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate medication satisfaction after at least 4 weeks of paliperidone ER (extended-release), an antipsychotic, treatment in patients with schizophrenia who were previously taking either 4 or 6 mg of risperidone daily by mouth, but who are not satisfied with their treatment.

DETAILED DESCRIPTION:
Paliperidone ER has been shown to be effective compared to placebo ("a sugar pill") in the acute treatment and maintenance of patients with schizophrenia. Paliperidone ER combines an active metabolite of another antipsychotic, risperidone, with manufacturing technology allowing more gradual release of the drug and less difference in high and low blood levels of the drug. Side effects to medications are sometimes due to wide differences in these high and low blood levels. Recent research has shown that many patients with schizophrenia discontinue their antipsychotic medication due to "subject-choice". Therefore, it is important that research studies attempt to measure patients' satisfaction with antipsychotic medication, in addition to measuring how they respond on tests of effectiveness. This study has been designed to evaluate antipsychotic medication satisfaction in patients who continue to have symptoms of schizophrenia, and who say they are dissatisfied with their current risperidone treatment. The primary outcome is the change in the Medication Satisfaction Questionnaire (MSQ) score, from baseline to the Week 6 endpoint. These patients are randomized (like flipping a coin) as to when their risperidone (4 mg to 6 mg per day) is switched to paliperidone ER. Because the study is 'blinded', neither the study doctor nor the patient will know when treatment with risperidone is stopped and treatment with paliperidone ER begins. Throughout the study all patients continue to receive antipsychotic medication daily. Patients will continue on the same daily dose of risperidone until their randomly assigned switch to paliperidone ER. All patients will be switched to paliperidone ER over the course of study and once switched continue to take paliperidone ER for the remainder of the study. Paliperidone ER is started at 6 mg/day and can be increased to 9 mg/day or 12 mg/day at the doctor's discretion. Effectiveness and safety will be measured at visits scheduled weekly for the first four weeks and then at the Week 6 endpoint. At each visit, patients will be asked to complete psychiatric tests and questionnaires that will measure effectiveness and patient satisfaction with the medicine. They will also complete tests and evaluations for safety, including electrocardiograms (ECGs, electrical tracings of the heart) and blood samples at the beginning and end of the study. Each patient receives two blinded capsules by mouth once daily in the morning for 6 weeks. Patients taking risperidone receive either a 4-mg or 6-mg capsule plus a placebo capsule. When patients are switched, Paliperidone ER is started at 6 mg/day the day after risperidone is discontinued and can be increased to 9 mg/day or 12 mg/day at the doctor's discretion. Paliperidone 3-mg and 6-mg capsules are combined with placebo to equal the total dose in two capsules.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand, in the opinion of the investigator, the informed consent form.
* be diagnosed with schizophrenia
* report dissatisfaction with current medication
* have an aspect of schizophrenia management which could potentially benefit from a change in antipsychotic medication
* receive risperidone 4 mg or 6 mg for at least 4 weeks before the start of the study.

Exclusion Criteria:

* Unable to swallow study drug whole with the aid of water
* cannot have received an investigational drug, used an investigational medical device, or participated in a clinical study that altered their medication within 6 months before the first administration of study drug, or have participated in more than 2 investigational drug studies within the past 12 months
* no other major mental health diagnosis except for tobacco dependance
* no use of cocaine or heroin within 3 months before the first administration
* no history of treatment with any antipsychotic in addition to treatment with risperidone, or treatment with paliperidone, within 30 days before the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (40):
- United States (15):
  - Cerritos, California
  - Garden Grove, California
  - Huntington Beach, California
  - Pico Rivera, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Flowood, Mississippi
  - Clementon, New Jersey
  - Brooklyn, New York
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Irving, Texas
- Argentina (7):
  - Miami, FL
  - Buenos Aires
  - Ciudad Autonoma de
  - Cordoba Crd
  - Mendoza
  - Mendoza Men
  - Rosario
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Bogotá S/N
  - Bucaramanga S/N
- Czechia (3):
  - Pilsen
  - Prague
  - Sternberk
- Slovakia (5):
  - Bojnice
  - Bratislava
  - Michalovce
  - Rimavská Sobota
  - Žilina
- Ukraine (6):
  - Dnipropetrovsk
  - Donetsk
  - Kiev
  - Lviv
  - Odesa
  - Village Stepanovka Kherson

REFERENCES:
- [Derived] Canuso CM, Grinspan A, Kalali A, Damaraju CV, Merriman U, Alphs L, Awad AG. Medication satisfaction in schizophrenia: a blinded-initiation study of paliperidone extended release in patients suboptimally responsive to risperidone. Int Clin Psychopharmacol. 2010 May;25(3):155-64. doi: 10.1097/YIC.0b013e3283372977. PMID 20216424
- See also: A blinded-initiation study of medication satisfaction in subjects with schizophrenia treated with paliperidone ER after suboptimal response to oral risperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=76&filename=CR014347_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- PALI ER Immediate Initiation: Subjects randomly assigned at the baseline visit to an immediate initiation of paliperidone ER from oral risperidone were to receive blinded paliperidone ER for a total of 6 weeks (Immediate Initiation group).
- PALI ER Delayed Initiation: Subjects randomly assigned to a delayed initiation were to receive blinded resperidone at their baseline dose of 4 or 6 mg for 2 weeks and were to be initiated on blinded paliperidone ER at Day 14 for 4 weeks (Delayed Initiation group).
Period: Randomized Population
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation
Started | 100 (Number of Subjects Randomized) | 101 (Number of Subjects Randomized)
Completed | 100 | 101
Not Completed | 0 | 0
Period: Safety Analysis Set
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation
Started | 100 | 101
Completed | 98 (Two patients were randomized but not treated.) | 99 (Two patients were randomized but not treated.)
Not Completed | 2 | 2
Not completed — Did Not Receive Study Medication | 2 | 2
Period: Intent-to-Treat (ITT) Analysis Set
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation
Started | 98 | 99
Completed | 95 (Patients who received at least one dose of study drug and have some follow-up efficacy data.) | 96 (Patients who received at least one dose of study drug and have some follow-up efficacy data.)
Not Completed | 3 | 3
Not completed — No Follow-up Efficacy Data | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- PALI ER Delayed Initiation: Subjects randomly assigned to a delayed initiation were to receive blinded resperidone at their baseline dose of 4 or 6 mg for 2 weeks and were then to be initiated on blinded paliperidone ER at Day 14 for 4 weeks (Delayed Initiation group).
- Total: Total of all reporting groups
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Analysis Set.
  years | 41.1 (12.5) | 40.2 (11.4) | 40.6 (11.9)
Sex/Gender, Customized [Number; unit: participants] — Safety Analysis Set.
  participants
    Male | 58 | 53 | 111
    Female | 40 | 46 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety Analysis Set.
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 31 | 26 | 57
    White | 61 | 69 | 130
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Medication Satisfaction Questionnaire (MSQ) Score Change From Baseline to the Week 6 Endpoint.
Description: The MSQ is a 7-point, verbally administered, Likert-type scale rated as follows: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied Nor Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Worst value is 1 (Extremely Dissatisfied) and best value is 7 (Extremely Satisfied).
Time Frame: Change from Baseline in MSQ Score at Week 6 Last Observation Carried Forward (LOCF)
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Groups:
- Overall: Combined subjects in the paliperidone ER Immediate Initiation and paliperidone ER Delayed Initiation groups.
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 95 | 96 | 191
Points on a scale | 2.5 (1.2) | 2.3 (1.5) | 2.4 (1.4)
Statistical Analysis 1: Comparison: Overall; Sample size for this study was based on changes in the MSQ scores within subjects from baseline to endpoint using a one-sample paired t-test. A sample size of 97 subjects was shown to have 90% power at endpoint to detect a mean change from baseline of 0.5 units on the MSQ score, with a standard deviation of 1.5. Allowing for extra variability from subjects with prior generic risperidone (instead of branded risperidone) use, this number was increased to 150 subjects; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value based on a paired t-test for a within-group comparison; Mean Difference (Final Values) = 2.4, Standard Deviation 1.4

2. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) Score Change From Baseline to Week 2 (Observed).
Description: as for outcome 1
Time Frame: Change from Baseline in MSQ Score at Week 2
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 93 | 95 | 188
Points on a scale | 2.0 (1.4) | 1.6 (1.4) | 1.8 (1.4)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = 1.8, Standard Deviation 1.4

3. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) Score Change From Baseline to Week 4 (Observed).
Description: as for outcome 1
Time Frame: Change from Baseline in MSQ Score at Week 4
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 89 | 91 | 180
Points on a scale | 2.4 (1.2) | 2.1 (1.5) | 2.3 (1.4)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 2.3, Standard Deviation 1.4

4. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) Score Change From Baseline to Week 6 (Observed).
Description: as for outcome 1
Time Frame: Change from Baseline in MSQ Score at Week 6
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 85 | 87 | 172
Points on a scale | 2.5 (1.2) | 2.4 (1.3) | 2.5 (1.3)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = 2.5, Standard Deviation 1.3

5. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) - Categorical Summary - Dichotomized Categories - Week 2 (Observed).
Description: as for outcome 1
Time Frame: Week 2
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Number; unit: Participants
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 93 | 95 | 188
Participants
  Satisfied (score 5-7) | 63 | 43 | 106
  Dissatisfied (score 1-4) | 30 | 52 | 82
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.002, Fisher Exact; P-values for the study group comparisons using dichotomized categories are based on Fisher's Exact Test

6. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) - Categorical Summary - Dichotomized Categories - Week 4 (Observed).
Description: as for outcome 1
Time Frame: Week 4
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Number; unit: Participants
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 89 | 91 | 180
Participants
  Satisfied (score 5-7) | 75 | 64 | 139
  Dissatisfied (score 1-4) | 14 | 27 | 41
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.033, Fisher Exact; P-values for the study group comparisons using dichotomized categories are based on Fisher's Exact Test

7. Other Pre Specified Outcome: Positive and Negative Syndrome Scale (PANSS) Total Score Change From Baseline to Week 6 Endpoint
Description: The PANSS is a 30-item scale designed to capture numerous symptoms of schizophrenia, including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale as follows: 1=Absent, 2=Minimal, 3=Mild,4=Moderate, 5=Moderate Severe, 6=Severe, 7=Extreme. This scale has been shown to be sensitive to changes associated with medication treatment. In addition to a total score, this assessment yields separate scores along a Positive Syndrome, a Negative Syndrome, and a General Psychopathology Scales. Worst value is 210, best value is 30.
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 95 | 96 | 191
Points on a scale | -13.5 (12.2) | -12.3 (14.0) | -12.9 (13.1)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = -12.9, Standard Deviation 13.1

8. Other Pre Specified Outcome: Clinical Global Impression - Severity (CGI-S) Change From Baseline to Week 6 Endpoint
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a subject. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill subjects". Worst value is 7 and best value is 1.
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 95 | 96 | 191
Points on a scale | -0.8 (0.9) | -0.8 (1.0) | -0.8 (0.9)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = -0.8, Standard Deviation 0.9

9. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) - Categorical Summary - Dichotomized Categories - Week 6 (Observed).
Description: as for outcome 1
Time Frame: Week 6
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Number; unit: Participants
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 85 | 87 | 172
Participants
  Satisfied (score 5-7) | 77 | 71 | 148
  Dissatisfied (score 1-4) | 8 | 16 | 24
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.123, Fisher Exact — P-values for the study group comparisons using dichotomized categories are based on Fisher's Exact Test

10. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) - Categorical Summary - Dichotomized Categories - Week 6 LOCF.
Description: as for outcome 1
Time Frame: Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Number; unit: Participants
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 95 | 96 | 191
Participants
  Satisfied (score 5-7) | 83 | 75 | 158
  Dissatisfied (score 1-4) | 12 | 21 | 33
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.125, Fisher Exact; P-values for the study group comparisons using dichotomized categories are based on Fisher's Exact Test

11. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Global Satisfaction Score Change From Baseline to the Week 6 Endpoint
Description: The TSQM is a 14-item subject-assessed evaluation of treatment medication including 4 factors, Effectiveness (items 1-3), Side Effects (items 4-8), Convenience (items 9-11)and Global Satisfaction (items 12-14). Item 14 states "taking all things into account, how satisfied or dissatisfied are you with this medication?" and utilizes the following responses on a 7-point Likert scale: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied Nor Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Worst value is 0 and best value is 100.
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 95 | 96 | 191
Points on a scale | 30.2 (22.6) | 26.4 (23.6) | 28.3 (23.1)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = 28.3, Standard Deviation 23.1

12. Secondary Outcome: Short Form-36 Health Survey (SF-36) Physical Health Composite Score Change From Baseline to the Week 6 Endpoint
Description: The SF-36 is a well-validated and widely used quality-of-life instrument employed in numerous disease states, including schizophrenia. It is a self-administered survey that measures eight domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Scoring of the SF-36 was based on the SF-36 Manual and Interpretation Guide. Worst value is 0 and best value is 100.
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 88 | 91 | 179
Scores on a scale | 0.8 (8.4) | 2.1 (6.4) | 1.5 (7.5)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = 1.5, Standard Deviation 7.5

13. Secondary Outcome: Short Form-36 Health Survey (SF-36) Mental Health Composite Score Change From Baseline to the Week 6 Endpoint
Description: as for outcome 12
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 88 | 91 | 179
Scores on a scale | 6.7 (10.3) | 7.2 (10.6) | 7.0 (10.4)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = 7.0, Standard Deviation 10.4

14. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Change From Baseline to the Week 6 Endpoint
Description: The PSQI is a 2-part questionnaire that assesses sleep quality and disturbances in seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each domain is rated on a 4-point scale as follows: 0=Not during the past month, 1=Less than once a week, 2=Once or twice a week, 3=Three or more times a week. Total scores range from zero to 21; increasing scores indicate poorer sleep quality and total scores greater than 5 suggest significant sleep disturbance.
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 84 | 84 | 168
Points on a scale | -2.3 (4.3) | -2.2 (4.4) | -2.3 (4.3)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = -2.3, Standard Deviation 4.3

15. Secondary Outcome: Modified COVI Anxiety Scale (m-COVI) Change From Baseline to the Week 6 Endpoint
Description: The standard COVI Anxiety Scale is an investigator-assessed measure of the severity of anxiety symptoms on 4 items: verbal report, behavior, somatic symptoms, and relationship to study drug. Each dimension is assessed in 5 to 10 minutes using a 5-point scale as follows: 1=Not at all, 2=Somewhat, 3=Moderately, 4=Considerably, to 5=Very much. For this study, the standard COVI Anxiety Scale was modified to improve psychometric properties by incorporating anchor points for symptom severity, frequency, and duration and for functional impairment. Worst value is 20 and best value is 4.
Time Frame: Change from Baseline to Week 6 LOCF
Population: Intent-to-Treat Population with non-missing values at this timepoint
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Number analyzed (Participants) | 88 | 80 | 168
Points on a scale | -1.4 (2.8) | -1.3 (3.2) | -1.3 (3.0)
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-value for within-group comparison based on a paired t-test; Mean Difference (Final Values) = -1.3, Standard Deviation 3.0

ADVERSE EVENTS:
Arm/Group | PALI ER Immediate Initiation | PALI ER Delayed Initiation | Overall
Serious Adverse Events (participants affected / at risk) | 3/98 | 4/99 | 7/197
Other Adverse Events (participants affected / at risk) | 49/98 | 56/99 | 105/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PALI ER Immediate Initiation (N=98) | PALI ER Delayed Initiation (N=99) | Overall (N=197)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Schizophrenia (Psychiatric disorders) | 2 | 4 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PALI ER Immediate Initiation (N=98) | PALI ER Delayed Initiation (N=99) | Overall (N=197)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 4 (4)
Hyperprolactinaemia (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 9 (9) | 15 (15)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 5 (6) | 8 (10)
Pancreatitus acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Salivary Hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Irritability (General disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 3 (4)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood prolactin increased (Investigations) | 3 (3) | 2 (2) | 5 (5)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 2 (2) | 3 (3) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Bradykinesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 6 (6)
Dizziness postural (Nervous system disorders) | 3 (3) | 3 (3) | 6 (6)
Dyskinesia (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Dystonia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 8 (9) | 7 (7) | 15 (16)
Hypertonia (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 3 (3) | 3 (3) | 6 (6)
Somnolence (Nervous system disorders) | 5 (5) | 8 (9) | 13 (14)
Tremor (Nervous system disorders) | 2 (2) | 3 (4) | 5 (6)
Abulia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 2 (5) | 3 (6)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 5 (5)
Delusion (Psychiatric disorders) | 0 (0) | 2 (3) | 2 (3)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 9 (10) | 9 (10) | 18 (20)
Libido decreased (Psychiatric disorders) | 2 (2) | 3 (3) | 5 (5)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 2 (3) | 4 (7) | 6 (10)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 3 (3)
Galactorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less